CLINICAL TRIAL: NCT06773702
Title: Valutazione Dell'attività Motoria Dello Sfintere Esofageo Superiore Nei Pazienti Con Sintomi Extra Esofagei Da Reflusso
Brief Title: Evaluation of Upper Esophageal Sphincter Motor Activity in Patients with Extra Esophageal Reflux Symptoms
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: VAM-SES-SEER2019
Record Dates: First submitted 2024-12-03; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-11

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with laryngopharyngeal reflux symptoms: Gastroenterological evaluation by esophageal manometry, 24-hour Ph impedance testing, Otolaryngological evaluation by laryngoscopy
  Interventions: Other: gastroenterology and otolaryngological evaluation

INTERVENTIONS:
Other: gastroenterology and otolaryngological evaluation — * Gastroenterology evaluation: presence and intensity of esophageal symptoms of gastro esophageal reflux disease, high-resolution esophageal manometry, and 24-hour pH-impedancometry in the absence of PPI therapy.
  * otolaryngological evaluation: presence and intensity of laryngopharyngeal reflux symptoms, laryngoscopy.

SUMMARY:
To evaluate the presence of motor changes of the upper esophageal sphincter detectable by high-resolution manometry in patients with oropharyngeal symptoms referable to extra-esophageal reflux manifestations.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a condition that occurs when the passage of gastric contents into the esophagus becomes clinically symptomatic and results in the appearance of complications. The incidence is higher in countries with high socioeconomic status; in fact, the prevalence in the US is estimated to be between 15 and 30 percent of the population compared with 5 to 10 percent in eastern countries such as China. 1 Typical manifestations are heartburn and acid regurgitation; however, in some cases it may manifest with extraesophageal symptoms, termed atypical, resulting from the involvement of anatomical areas of otolaryngological and pulmonary relevance.

According to the 2006 Montreal classification (Figure 1), still the reference of gastroesophageal reflux disease, the disease can manifest with:

1. esophageal syndrome, subdivided into:

   * symptomatic, without esophageal injury (typical reflux syndrome, Chest pain syndrome)
   * syndrome with esophageal damage (esophagitis, stenosis, Barrett's esophagus and Adenocarcinoma of the esophagus)
2. extraesophageal syndrome, subdivided into:

   * association with established reflux disease (chronic cough, laryngitis, asthma, dental erosions)
   * association with proposed reflux disease (pharyngitis, sinusitis, idiopathic pulmonary fibrosis, recurrent otitis media).

A study performed by Francis DO in the United States in 2013 showed how the management of extra esophageal reflux disease substantially burdens public spending. In fact, it was found that the cost for the first year of evaluation and treatment of patients presenting with extra esophageal reflux symptoms is five times higher than the management of typical esophageal reflux disease. The cause of this discrepancy is precisely the absence of a definitive diagnosis and standard treatment, which result in difficult management of the disease.

While there is ample literature regarding the association between MRGE and alteration of the lower esophageal sphincter, little is described about the correlation between alterations in pharyngo-laryngeal motor activity and the upper esophageal sphincter in patients with extraesophageal reflux disease symptoms.

Indeed, it is hypothesized that the reflux of acidic material at the level of the larynx may be due to a dysfunction of the sphincter that acts as an escape valve between the esophagus and pharyngo-larynx. With the development of high-resolution manometry, which, unlike conventional manometry, has no spatial gaps and allows for a faithful representation of esophageal motor function in time and space, a detailed study of oropharyngeal and upper esophageal sphincter motor activity can be achieved

The observational, non-interventional nature of the study is based on two main elements:

1. the evaluation of data obtained from high-resolution esophageal manometry in patients with extra-esophageal reflux symptoms
2. the comparison of data obtained from high-resolution esophageal manometry with 24-hour PH-impedancemetry and otolaryngological scores of laryngopharyngeal reflux (Reflux symptom Index, Reflux Finding Score) Patients participating in the study will not undergo any procedures beyond normal daily clinical practice; likewise, the clinical variables that will be collected for the study are those that are commonly collected by the physician in daily clinical practice.

ELIGIBILITY:
Inclusion criteria.

* Age between 18 and 80 years.
* Patients with laryngopharyngeal reflux symptoms.
* Obtaining informed consent. Exclusion criteria.
* Patients with tobacco habit.
* Patients with occupational exposure to irritants (artisans and industrial workers).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All referral patients to the Gastrointestinal Functional Exploration outpatient clinic with symptoms of laryngo-pharyngeal reflux who need to have gastroenterologic evaluation by esophageal manometry, 24-hour Ph impedance testing, and ENT evaluation by laryngoscopy and who meet the inclusion criteria will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the presence of motor changes of the upper esophageal sphincter detectable on high-resolution manometry in patients with oropharyngeal symptoms referable to extra-esophageal reflux manifestations. | 1 year
  Evaluate the presence of motor changes of the upper esophageal sphincter detectable on high-resolution manometry in patients with oropharyngeal symptoms referable to extra-esophageal reflux manifestations.

SECONDARY OUTCOMES:
PH-impedancemetry | 1 year
  The secondary objectives of the study are contingent on the actual presence of manometric alterations of the upper esophageal sphincter in patients with extraesophageal syndrome. Basically, if no manometric changes are present, secondary objectives will: assess the association between manometric changes and the result of PH-impedancemetry
Reflux Index Score | 1 year
  The secondary objectives of the study are contingent on the actual presence of manometric alterations of the upper esophageal sphincter in patients with extraesophageal syndrome. Basically, if no manometric changes are present, secondary objectives will: evaluate the association between manometric alterations and the result of Reflux Index Score
Reflux Symptom Index | 1 year
  The secondary objectives of the study are contingent on the actual presence of manometric alterations of the upper esophageal sphincter in patients with extraesophageal syndrome. Basically, if no manometric changes are present, secondary objectives will: evaluate the association between manometric alterations and the result of the Reflux Symptom Index

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Torresan, MD, Principal Investigator — IRCCS AOUBo
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No